CLINICAL TRIAL: NCT06991725
Title: Botulinum Neurotoxin for Children With Cerebral Palsy: a Delicate Balance Between Clinical Benefits and Muscular Harm
Brief Title: Botulinum Neurotoxin for Children With CP: a Delicate Balance Between Clinical Benefits and Muscular Harm
Acronym: Bo-Balance
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62187_Bo-Balance
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: Spastic Cerebral Palsy; Muscle composition; 3D freehand ultrasound; Shear wave elastography; Muscle morphology; Range of motion; Stiffness; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with spastic cerebral palsy: Children between 2 years and 16 years old
- Typically developing children: Children between 2 years and 16 years old

SUMMARY:
A cross-sectional design study will be carried out to explore the morphological muscle properties and alterations in muscle composition on a macroscopic level in children with spastic cerebral palsy (CP). Muscle composition will be assessed using quantitative Magnetic Resonance Imaging (qMRI) and shear wave elastography (SWE), while macroscopic muscle size properties will be evaluated through 'Three-dimensional freehand ultrasound (3DfUS).

DETAILED DESCRIPTION:
Background: Altered muscle composition, including increased fat infiltration and collagen content, is a key factor in impaired muscle function in cerebral palsy (CP). However, quantitative data on muscle composition in CP is limited. Traditional methods like ultrasound can only indirectly assess these changes through echo-intensity, while invasive muscle biopsies are impractical for children. Recent advancements in quantitative Magnetic Resonance Imaging (qMRI) and shear wave elastography (SWE) provide non-invasive alternatives. The qMRI Dixon sequence can assess fat infiltration, while the T1ρ sequence can estimate collagen content. SWE can measure passive muscle stiffness as a surrogate marker for collagen. Combining these techniques allows for a comprehensive evaluation of muscle composition and its impact on muscle function in CP. Next to muscle composition, children with CP also exhibit muscle size deficits compared to typically developing (TD) children. More specifically, when accounting for the effect of natural muscle growth, normalized muscle volume was found to be reduced, which could be attributed to a reduction in normalized cross-sectional area and normalized muscle belly length. Because muscle morphology (or muscle size) can be estimated using accessible ultrasonography techniques, alterations in muscle size have been well-described in growing children with CP. However, since muscle composition can only be estimated through more advanced, recent muscle imaging techniques, its alteration in CP remains underexplored.

Aim: To comprehensively describe the alterations in intrinsic muscle properties, the evaluation of altered muscle morphology (or muscle size) will be complemented with the description of alterations in muscle composition. Unlike muscle size, which increases with age, muscle composition remains relatively stable in typically developing children. Since comprehensive assessment of muscle composition requires MRI, a less practical tool compared to ultrasonography, the study will adopt a cross-sectional descriptive design. We aim to create an integrated dataset of muscle composition combined with muscle size, passive muscle stiffness and clinical assessments for CP and TD children that are equally distributed over pre-school, grade-school and teen-aged.

Methods/design: Children with CP who participated in previous studies within this project will be invited to join the current study. 34 children with CP participants will be recruited to reach the target sample size . The CP group will be evenly divided between those who are botulinum neurotoxin (BTX) naïve and those who have received BTX treatment. Only children with a Gross Motor Function Classification System (GMFCS) level of I, II, or III will be included. In total, 34 children with CP and 17 age-matched typically developing (TD) children will be enrolled in the study.

Participants will be evaluated at the University Hospitals Leuven (UZ Leuven) at campus Gasthuisberg or campus Pellenberg. Data will be collected during a hospital visit and every participant will undergo at least a 3DfUS and SWE measurement of the medial gastrocnemius. Other information that will be collected out of the available medical records includes the results of the structural brain MRI, the use of medication, treatment details (physiotherapy, orthotics and/or orthopedic interventions), anthropometric measures (body weight and length and leg lengths), data of a standard clinical examination (joint range of motion, spasticity, and muscle selectivity and strength).

ELIGIBILITY:
- Children with spastic cerebral palsy

Inclusion criteria:

* Children (boys/girls) with congenital brain lesion, confirmed with neuro-imaging such as MRI
* At high-risk for CP or diagnosed spastic type of CP
* (Suspected) Gross Motor Function Classification Scale (GMFCS) Level I-III
* Uni or bilateral involvement
* Aged between 2-16 years

Exclusion criteria:

* Presence of dyskinesia or ataxia
* Severe co-morbidities (cognitive problems)
* BTX treatment in past 10 months
* Previous surgery less than 12 months at the investigated muscles.
* Previous orthopedic or neurosurgery
* Severe ankle deformities
* Weight for height values >2SD from mean

  * Typically developing children

Inclusion criteria:

• Aged between 2-16 years

Exclusion criteria:

* History of neurological, orthopedic or muscular problems
* Involvement in an elite or high-performance sporting program (Children performing the same sports for > 5 hours/week will be excluded)

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic cerebral palsy, who have routine follow-up care at the CP reference center of the University Hospitals Leuven. Typically developing children are recruited through the social (family and friends) and professional (colleagues) network of involved researchers and thesis students, who approach participants through flyers, social media.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the muscle volume of the medial gastrocnemius muscle | Cross-sectional data collection at day 1.
  Estimation of the muscle belly volume by 3DfUS. Muscle volume will be normalized to anthropometric growth.
Evaluation of the muscle length of the medial gastrocnemius muscle | Cross-sectional data collection at day 1.
  Estimation of the muscle belly length, tendon length and muscle tendon unit complex length by 3DfUS. Muscle lengths will be normalized to anthropometric growth
Evaluation of the muscle echo-intensity of the medial gastrocnemius muscle | Cross-sectional data collection at day 1.
  Estimation of the echo-intensity by 3DfUS.
Evaluation of the fat fraction of the medial gastrocnemius muscle. | Cross-sectional data collection at day 1.
  Estimation of the fat fraction by Dixon sequence (MRI): a comparison of muscle fat fraction between children with CP and healthy age-matched TD controls in different age groups.
Indirect evaluation of collagen content of the medial gastrocnemius muscle | Cross-sectional data collection at day 1.
  Indirect estimation of collagen content by T1ƿ relaxation time (MRI): a comparison between children with CP and healthy age-matched TD controls in different age groups.
Evaluation of passive muscle stiffness across the medial gastrocnemius muscle. | Cross-sectional data collection at day 1.
  Estimation of the passive muscle stiffness by shear modulus (SWE): a comparison of passive muscle stiffness between children with CP and healthy age-matched TD controls in different age groups.
Evaluation of differences in fat fraction in different regions across the medial gastrocnemius muscle. | Cross-sectional data collection at day 1.
  Comparison of differences in fat fraction across three regions (proximal, midbelly, distal) of the muscle belly in children with CP compared to TD children.
Evaluation of differences in passive muscle stiffness in different regions across the medial gastrocnemius muscle. | Cross-sectional data collection at day 1.
  Comparison of differences in passive muscle stiffness across three regions (midbelly, distal, upper fascia of midbelly) of the muscle belly in children with CP compared to TD children.
Evaluation of the muscle strength (ankle torque). | Cross-sectional data collection at day 1.
  Evaluating the muscle strength (ankle torque) using the handheld dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof.dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium